CLINICAL TRIAL: NCT04740476
Title: An Open-Label Extension Study for Patients With Dravet Syndrome Who Previously Participated in Studies of STK-001
Brief Title: An Open-Label Extension Study of STK-001 for Patients With Dravet Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stoke Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STK-001-DS-501
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Dravet Syndrome
Keywords: Pediatric epilepsy; Epileptic Encephalopathies; Refractory Myoclonic Epilepsy; Severe Myoclonic Epilepsy in Infancy
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- zorevunersen (STK-001) multiple dose levels (Experimental): Enrollment of patients after completion of Study STK-001-DS-101 or Study STK-001-DS-102 if eligible. Patients will receive IT administration of study drug zorevunersen at the dose level they received while participating in Study STK-001-DS-101 or STK-001-DS-102, or at a dose level recommended by the Safety Monitoring Committee (SMC).The highest dose administered in this study may not exceed that which has already been evaluated in an zorevunersen Phase 1/2 study, and doses above 45 mg/dose in this study require approval from the Food and Drug Administration (FDA). Patients will initially receive 3 doses, one every approximately 4 months (16 weeks). Patients who are tolerating treatment may continue treatment with doses approximately every 4 months, with an End of Study/Follow-up Visit 24 weeks after the last dose of study drug. Patients who do not continue treatment after the third dose will have a Follow-up Visit (V5) at Week 48 and an End of Study Visit at Week 56.
  Interventions: Drug: zorevunersen (STK-001)

INTERVENTIONS:
Drug: zorevunersen (STK-001) — zorevunersen drug product is an antisense oligonucleotide administered as an intrathecal injection.

SUMMARY:
Stoke Therapeutics is evaluating the long-term safety & tolerability of repeated doses of zorevunersen (STK-001) in patients with Dravet syndrome who previously participated in studies of zorevunersen. Change in seizure frequency and overall clinical status, and quality of life will be measured as secondary endpoints in this open-label study.

DETAILED DESCRIPTION:
This study is a multi-center, open-label, multiple-dose, safety extension study for patients who have completed another study of zorevunersen and meet study eligibility criteria. zorevunersen is an investigational new medicine for the treatment of Dravet syndrome. Zorevunersen is an antisense oligonucleotide (ASO) that is intended to increase the level of productive SCN1A messenger RNA (mRNA) and consequently increase the expression of the sodium channel Nav1.1 protein. This RNA-based approach is not gene therapy, but rather RNA modulation, as it does not manipulate nor insert genetic deoxyribonucleic acid (DNA).

Zorevunersen is designed to upregulate Nav1.1 protein expression from the nonmutant (wild-type) copy of the SCN1A gene to restore physiological Nav1.1 levels. Nav1.1 levels are reduced in people with Dravet syndrome. Stoke has generated preclinical data demonstrating proof-of-mechanism for zorevunersen.

ELIGIBILITY:
Inclusion Criteria:

* Completed dosing with zorevunersen and the End of Study Visit in Study STK-001-DS-101 or Study STK-001-DS-102, with an acceptable safety profile per Investigator judgment.
* Had satisfactory compliance with study visits and procedures in Study STK-001-DS-101 or Study STK-001-DS-102 per Investigator and Sponsor judgment.
* Completed Study STK-001-DS-101 or STK-001-DS-102 within 4 weeks of the start of their participation in Study STK-001-DS-501 unless approved by sponsor.

Exclusion Criteria:

* Met any withdrawal criteria from Study STK-001-DS-101 or STK-001-DS-102.
* Currently treated with an antiepileptic drug (AED) acting primarily as a sodium channel blocker, as maintenance therapy, including phenytoin, carbamazepine, oxcarbazepine, lamotrigine, lacosamide or rufinamide (with the exception of cenobamate, which is permitted).
* Clinically significant unstable medical conditions other than epilepsy.
* Clinically relevant symptoms or a clinically significant illness (in the judgment of the Investigator) at Screening or prior to dosing on Day 1, other than epilepsy.
* Spinal deformity or other condition that may alter the free flow of CSF or has an implanted CSF drainage shunt.
* Treated (or is being treated) with an investigational product (other than zorevunersen) since participating in Study STK-001-DS-101 or STK-001-DS-102.
* Participating in an observational study, they are excluded unless approved by the Sponsor.

Min Age: 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety of multiple doses of zorevunersen | Screening (Day -1) until 6 months after multiple drug dosing
  Safety variables for analysis include the incidence, type, severity, and seriousness of AEs, and changes in vital signs, ECG, laboratory, immunogenicity, physical examination, and outcomes on the cerebellar function clinical screening battery.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameters | Dosing (Day 1) until 6 months after multiple drug dosing
  Analysis of plasma concentrations of zorevunersen
Exposure of zorevunersen in Cerebrospinal Fluid (CSF) | Dosing (Day 1) and every 4 months until last study drug dosing day
  Measurement of zorevunersen concentrations
Measurement of Seizure Frequency | Screening (Day -1) until 6 months after multiple drug dosing
  Measurement of Seizure Frequency (by paper diary)
Change in overall clinical status | Screening (Day -1) until 6 months after multiple drug dosing
  Change in overall clinical status as measured by the Clinical Global Impression of Change (CGIC) and the Caregiver Global Impression of Change (CaGIC)
Change in Quality of Life | Screening (Day -1) until 6 months after multiple drug dosing
  Change in quality of life as measured by the EuroQoL-five dimensions, youth version (EQ-5D-Y) instrument

CONTACTS AND LOCATIONS:
Overall Officials: Ann Dandurand, MD, Study Director — Medical Director
Locations (17):
- United States (17):
  - University of California San Francisco Medical Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Florida Hospital for Children, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Comprehensive Epilepsy Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT LeBonheur Pediatric Specialists, Inc., Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington